CLINICAL TRIAL: NCT05198128
Title: Ovarian Hyper Stimulation Syndrome Using Calcium Infusion
Brief Title: Ovarian Hyperstimulation Syndrome Using Calcium Infusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Said Ali, DR: ahmedsaidali, MCS CANDIDIATE, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2217-2021
Record Dates: First submitted 2021-12-19; First posted 2022-01-20 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: OHSS; calcium infusion; IVF; ICSI
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Calcium for Prevention of Ovarian Hyperstimulation Syndrome (OHSS)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium intravenous infusion (Experimental): intravenous infusion of 10 % calcium gluconate 10 mL in 200 mL of physiologic saline on the day of ovum pickup, day 1,day 2, and day 3 after ovum pickup were administered in study group.
  Intravenous infusion was performed within 30 minutes
  Interventions: Drug: Calcium intravenous infsuion
- saline (Placebo Comparator): 0.9 % saline intravenous infusion
  Interventions: Drug: 0.9 % saline

INTERVENTIONS:
Drug: Calcium intravenous infsuion — intravenous infusion of 10 % calcium gluconate 10 mL in 200 mL of physiologic saline on the day of ovum pickup, day 1,day 2, and day 3 after ovum pickup were administered in study group.
  Intravenous infusion was performed within 30 minutes
  Arms: Calcium intravenous infusion
Drug: 0.9 % saline — 0.9 % saline
  Arms: saline

SUMMARY:
the incidence of OHSS and clinical outcomes after calcium IV infusion in high-risk women undergoing ART

DETAILED DESCRIPTION:
Among assisted reproductive technologies (ART), ovarian hyperstimulation syndrome (OHSS) is a serious iatrogenic complication affects up to 30% of women undergoing ART and caries high risks of morbidity and mortality. Women with age younger than 35 years, those with history of polycystic ovary syndrome (PCOS), or having a history of previous OHSS are more susceptible to develop OHSS

ELIGIBILITY:
Inclusion Criteria:

- infertile women aged 20 to 38 years. BMI ranged from 18 to 40. serum FSH within normal limits( 1-12IU /l) presented with ovarian response suggestive of being at risk of developing OHSS because of the presence of at least 15 follicles of 10 mm or greater on the day of hCG administration.

Exclusion Criteria:

* endocrinopathies. a systemic disease. and Insulin-dependent diabetes Thyroid disease using any medication (e.g., insulin-sensitizing drugs and GnRH antagonists. patients need coasting for high risk of OHSS. patients need cycle cancellation. severe male infertility requiring testicular sperm extraction.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women undergoing Ovarian Hyperstimulation Syndrome
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-04-25 (Estimated); Study Completion 2023-05-10 (Estimated)

PRIMARY OUTCOMES:
OHSS rate | one year
  ovarain hyperstimulation syndrome

IPD SHARING:
Plan to Share IPD: No
not yet